CLINICAL TRIAL: NCT00839540
Title: Comparison of Candida Eradication and Serum Cidal Activity of Echinocandins in Patients With Presumptive Candidemia
Brief Title: Comparison of Candida Eradication and Serum Cidal Activity of Echinocandins
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gary E. Stein, Pharm.D. (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Gary E. Stein, Pharm.D., Professor of Medicine, Michigan State University
Organization: Michigan State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA-07-004
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Candidemia
Keywords: candidemia; echinocandin; micafungin; caspofungin
MeSH Terms: conditions — Candidemia | interventions — Micafungin; Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- micafungin 100 (Active Comparator): Patients receive Micafungin 100 mg qd
  Interventions: Drug: micafungin
- micafungin 200 (Active Comparator): Patients receive 200 mg Micafungin qd
  Interventions: Drug: Micafungin
- Caspofungin (Active Comparator): Patients receive caspofungin 70 mg LD followed by 50 mg qd
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: micafungin — 100 mg qd by slow IV infusion for 24 h
  Other Names: Micamine
  Arms: micafungin 100
Drug: Micafungin — 200 mg qd by slow IV infusion for 24 h
  Other Names: Micamine
  Arms: micafungin 200
Drug: Caspofungin — 70 mg LD followed by 50 mg qd by slow IV infusion for 24 h
  Other Names: Cancidas
  Arms: Caspofungin

SUMMARY:
The purpose of this pharmacokinetic (PK) and pharmacodynamic (PD) study is:

To study the rate and duration of serum cidal activity of caspofungin (CFG) and micafungin (MFG) against Candida isolates from the subject and against Candida glabrata with varying degrees of caspofungin susceptibilities.

This investigation will provide clinicians information supporting the use of caspofungin and micafungin in situations where Candida strains may be a cause of infection.

DETAILED DESCRIPTION:
Methods:

Patients - Adult patients with presumptive candidemia. Patients with severe neutropenia (<500) APACHE II scores > 20, or significant liver disease will be excluded. All will give written informed consent (Pappas et al. CID. Oct 1, 2007).

Drugs - Patients will receive either CFG: 70 mg loading dose (LD) followed by 50 mg once daily (qd) (8 patients), MFG: 100 mg qd (8 patients) or MFG: 200 mg qd (8 patients). All agents will be given by slow IV infusion (MFG will be supplied by Astellas).

Sera - Blood samples will be collected at the end of the infusion (peak) and at 12 h and 24 h (trough) after the beginning of an infusion (day 3-4).

Each patients sera will be tested (MIC and cidal activity) against their own Candida isolate (if isolated). In addition, recent clinical isolates of C. glabrata will also be tested against patient sera (time-kill) to verify previous in vitro and animal PD studies (Cota. AAC. Nov. 2006; Wiederhold. AAC. May 2007).

Results:

* Patient outcome, including Candida eradication, will be documented for each patient by repeat culture.
* Serum concentrations (lab to be determined) and PK analysis of each echinocandin will be determined for each patient.
* Serum cidal titers will be measured against each of the Candida isolates for each agent at each time period. Median and geometric mean Peak and duration of cidal activity will then be determined and compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with presumptive candidemia

Exclusion Criteria:

* Patients with severe neutropenia (<500)
* Patients with APACHE II scores > 20
* Patients with severe liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Stein, Pharm.D., Principal Investigator — Michigan State University
Locations (1):
- Sparrow Hospital, Lansing, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were inpatients (Sparrow Hospital) with probable fungal infections that required treatment with an antifungal; referral base was infectious disease consultations. The first subject was enrolled 12/24/08, with the last subject enrolled on 1/15/10.
Groups:
- Micafungin (M) 100: Patients receive Micafungin (M) 100 mg once daily (qd)
- Micafungin (M) 200: Patients receive 200 mg Micafungin (M) once daily
- Caspofungin (C) 50: Patients receive caspofungin 70 mg loading dose (LD) followed by 50 mg once daily (qd)
Period: Overall Study
Arm/Group | Micafungin (M) 100 | Micafungin (M) 200 | Caspofungin (C) 50
Started | 8 | 8 | 5
Completed | 8 | 8 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micafungin (M) 100 | Micafungin (M) 200 | Caspofungin (C) 50 | Total
Number analyzed (Participants) | 8 | 8 | 5 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 4 | 11
  >=65 years | 5 | 4 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.62 (16.13282) | 57.81 (17.38585) | 44.0 (20.43282) | 57.6 (18.65374)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 3 | 10
  Male | 6 | 3 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: Serum Cidal Activity as Tested Against Various Candida Isolates and Reported as Ex-vivo Effect (Log Inhibition of Growth)
Description: Serum cidal activity of serum collected at different timepoints from the patients will be tested against various Candida isolates and the ex-vivo effect reported as log inhibition (logrithmic measurement of the decrease in microbiological growth).
  These Candida isolates had a range of minimum inhibitory concentrations (MIC) to Caspofungin (C) and Micafungin (M).
Time Frame: Pre-treatment, 1.5 hour (h), 12 h and 24 h after receiving the drug
Population: Each subject received drug and had serum samples drawn at pre-treatment, 1.5h, 12h, and 24h after dosing.
Measure: Number; unit: Log inhibition
Units Other Than Participants: blood samples
Groups:
- Log Inhibition of 50 mg/Day Caspofungin on Candida Spp.: Measurement of the decrease in organism(Candida spp.) colony counts following exposure of serum containing Caspofungin based on 50 mg/day dosing, measured as Ex-vivo effect.
- Log Inhibition of 100 mg/Day Micafungin on Candida Spp.: Measurement of the decrease in organism(Candida spp.) colony counts following exposure of serum containing Micafungin based on 100 mg/day dosing, measured as Ex-vivo effect.
- Log Inhibition of 200 mg/Day Micafungin on Candida Spp.: Measurement of the decrease in organism(Candida spp.) colony counts following exposure of serum containing Micafungin based on 200 mg/day dosing, measured as Ex-vivo effect.
Arm/Group | Log Inhibition of 50 mg/Day Caspofungin on Candida Spp. | Log Inhibition of 100 mg/Day Micafungin on Candida Spp. | Log Inhibition of 200 mg/Day Micafungin on Candida Spp.
Number analyzed (Participants) | 5 | 8 | 8
Number analyzed (blood samples) | 10 | 19 | 19
Log inhibition
  C. albicans MIC: C, M 0.016 mg/L | 3 (NA) | 0.5 | 0
  C. glabrata MIC: C, M 0.06 mg/L | 3 (NA) | 1.5 | 0.5
  C. glabrata MIC: C, M 0.25 mg/L | 0.5 (NA) | 1 | 0.5
  C. albicans 119 FKS mutant MIC:C 1, M 0.16 mg/L | 0.5 | 0.5 | 1.5
  C. albicans 90 FKS mutant MIC: C 1, M 0.25 mg/L | 0 | 0.5 | 2
  C. albicans A-15 FKS mutant MIC: C 2, M0.5 mg/L | 0 | 0 | 0
  C. glabrata MIC: C 2, M 0.5 mg/L | 0 | 0 | 0
  C. albicans 117 FKS mutant MIC: C 8, M 0.83 mg/L | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Micafungin (M) 100 | Micafungin (M) 200 | Caspofungin (C) 50
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micafungin (M) 100 (N=8) | Micafungin (M) 200 (N=8) | Caspofungin (C) 50 (N=5)
Death (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) — Death due to disease progression (fungal infection), not related to study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No